CLINICAL TRIAL: NCT01873170
Title: Quantification of Immune Cells in Women Using Contraception
Brief Title: Quantification of Immune Cells in Women Using Contraception (CHIC II)
Acronym: CHIC-II
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sharon Achilles, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY19100126
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: HIV; Immune Cells (Mucosal and Systemic); Contraception
Keywords: immune cells; contraception; intrauterine device; IUD; copper; microflora; DMPA; etonogestrel; subdermal implant
MeSH Terms: interventions — Levonorgestrel; Ethinyl Estradiol-Norgestrel Combination; N,N-dimethyl-4-anisidine; Medroxyprogesterone Acetate; etonogestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma archive, vaginal swabs, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Combined Oral Contraceptive pills: Levonorgestrel/ethinyl estradiol 0.15mg/30mcg daily oral tabs x21 then 7 inert tabs
  Interventions: Drug: levonorgestrel exposure
- depot medroxyprogesterone acetate: 150mg DMPA intramuscular injection once every 3 months
  Interventions: Drug: DMPA exposure
- Levonorgestrel-intrauterine device: 52mg levonorgestrel intrauterine device
  Interventions: Drug: levonorgestrel exposure; Device: IUD insertion
- Copper intrauterine device: Copper T380A intrauterine device
  Interventions: Device: IUD insertion
- Etonogestrel contraceptive implant: 68mg etonogestrel subdermal implant
  Interventions: Drug: etonogestrel exposure; Device: subdermal contraceptive implant insertion
- Control: Low risk of pregnancy due to sterilization, heterosexual abstinence, or consistent condom use

INTERVENTIONS:
Drug: levonorgestrel exposure
  Other Names: LNG-IUD (Mirena); LNG/EE oral contraceptive pills (Levora)
  Groups: Combined Oral Contraceptive pills; Levonorgestrel-intrauterine device
Drug: DMPA exposure
  Other Names: DMPA (Depo-Provera 150mg IM)
  Groups: depot medroxyprogesterone acetate
Drug: etonogestrel exposure
  Other Names: ENG-implant (Nexplanon or Implanon)
  Groups: Etonogestrel contraceptive implant
Device: IUD insertion
  Other Names: LNG-IUD (Mirena); Copper T-380A IUD (ParaGard)
  Groups: Copper intrauterine device; Levonorgestrel-intrauterine device
Device: subdermal contraceptive implant insertion
  Other Names: ENG-implant (Nexplanon or Implanon)
  Groups: Etonogestrel contraceptive implant

SUMMARY:
This study is being done to understand if using birth control causes changes in the immune cells within the reproductive tract (including the cervix and the lining of the uterus) of healthy women. Immune cells are important because they help prevent infections from starting and help fight infections that have started. Immune cells are also the type of cells that HIV (human immunodeficiency virus) infects so understanding more about them will help to better understand how to prevent the spread of HIV.

Immune cells will be studied from the reproductive tract of women who want to start using one of the following contraceptives: an oral contraceptive pill (COC), Depo-Provera (DMPA), the levonorgestrel IUD (Mirena®), the copper IUD (ParaGard®), or the etonogestrel subdermal implant (Nexplanon®).Immune cells will also be studied from the reproductive tract of women who are not using birth control and who are not at risk of pregnancy for comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 34 years (inclusive) at screening
2. Non-pregnant women in general good health as determined by the site clinician
3. Premenopausal with history of regular menstrual cycles (regular cycles defined as occurring every 21-35 days when not using hormones and with a variation of typical cycle length of no more than 5 days)
4. Women enrolling into the control group only: Regular and consistent condom use, prior surgical sterilization by participant or sexual partner, or heterosexually abstinent for entire study participation
5. Able and willing to provide written informed consent to be screened for and to take part in the study. Including willingness to undergo all study-related assessments and follow all study-related procedures
6. Able and willing to provide adequate locator information
7. HIV-uninfected based on testing performed by study staff at screening (per HIV testing algorithm in Appendices I)
8. At screening and enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products while enrolled in this trial

Exclusion Criteria:

1. Use of any hormonal or intrauterine contraceptive method within 30 days of enrollment
2. Use of DMPA within 10 months of enrollment
3. Pregnancy or breastfeeding within 60 days of enrollment
4. Surgical procedure involving the pelvis in the 30 days prior to enrollment (includes dilation and curettage, cryosurgery and biopsy of the vagina, vulva, cervix, and endometrium)
5. Internal vaginal use of any device (includes sex toys, cervical caps, diaphragms, menstrual collection devices, and pessaries; excludes tampons and condoms) or product (includes N9, microbicide, douche, antifungal, steroid, or hormone) in the 30 days prior to enrollment
6. New sexual partner within 90 days of enrollment
7. Urogenital infection or suspected infection within 30 days of enrollment including: symptomatic candidiasis, trichomonas vaginalis, and symptomatic bacterial vaginosis; or cervical infection, including N. gonorrhea, C. trachomatis, or mucopurulent cervicitis; syphilis; HSV lesions, or other sores (Note: seropositive HSV without active lesions will not be excluded); acute pelvic inflammatory disease; urinary tract infection; recent exposure to a partner with GC, CT, Trichomonas, syphilis, or NGU
8. Any history of immunosuppression (includes diabetes, HIV infection, and chronic steroid use)
9. Antibiotic or antifungal therapy (vaginal or systemic) within 30 days of enrollment
10. Menses or other vaginal bleeding at the time of Enrollment* (*Women who have vaginal bleeding at the scheduled Enrollment Visit may return at a different date to be re-examined and possibly enrolled provided they are still within the 90-day screening window and meet all criteria).
11. Vaginal or anal intercourse within 36 hours prior to enrollment
12. Heterosexual intercourse since last menses that places the participant at risk of pregnancy (without condom use or sterilization of at least one partner)
13. History of hysterectomy
14. History of malignancy within the pelvis (includes uterus, cervix, vagina, and vulva)
15. Contraindication, allergy or intolerance to use of the contraceptive desired by the participant
16. Any condition that, in the opinion of the Investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women, age 18-34 years, who are HIV negative and non-pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Quantification and characterization of immune cell populations and HIV-tropic receptor expression | up to 6 months
  To quantify and characterize immune cell populations and HIV-tropic receptor expression in the upper and lower genital tract and blood at baseline and after 3 and 6 months of typical contraceptive use

SECONDARY OUTCOMES:
Assessing changes in the vaginal microflora within the first 6 months of contraceptive use | baseline, 3 months, 6 months
  To describe the microflora of the upper and lower genital tracts of healthy asymptomatic women before and after 3 and 6 months of typical contraceptive use and to assess changes in the vaginal ecology within the first 6 months of contraceptive use.

OTHER OUTCOMES:
Reproductive tract Microenvironment | baseline, 3 months, 6 months
  To assess if changes in the upper and lower genital tract microflora are correlated with alterations in immune cell populations

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Chen, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Center for Family Planning Research, Pittsburgh, Pennsylvania, United States